CLINICAL TRIAL: NCT03280004
Title: Reason Evaluation of Initial Treatment Failure in Patients With Community Acquired Pneumonia
Brief Title: Reason Evaluation of Initial Treatment Failure in Patients With CAP
Acronym: RECAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jun Xu, Dr, Peking Union Medical College Hospital
Other Study IDs: HS-1279
Record Dates: First submitted 2017-09-10; First posted 2017-09-12 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Moxifloxacin; Sodium Chloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Moxifloxacin group
  Interventions: Drug: Moxifloxacin Hydrochloride and Sodium Chloride Injection
- β-lactams group

INTERVENTIONS:
Drug: Moxifloxacin Hydrochloride and Sodium Chloride Injection — Moxifloxacin group will be given Moxifloxacin Hydrochloride and Sodium Chloride Injection and β-lactams group will be given β-lactam antibiotics for injection +/- Azithromycin for Injection.
  Groups: Moxifloxacin group

SUMMARY:
This research is to evaluate the effect of different antibiotics (Moxifloxacin Hydrochloride and Sodium Chloride Injection vs. β-lactam antibiotics for injection +/- Azithromycin for Injection) on the early deterioration or progression (<72 h of treatment) of community acquired pneumonia and to study the effect of the early deterioration or progression on the prognosis of community acquired pneumonia.

ELIGIBILITY:
Inclusion Criteria:

1. Age>=18y.
2. Diagnosed with CAP.
3. Need hospitalization.
4. Receive Moxifloxacin Hydrochloride and Sodium Chloride Injection or β-lactam antibiotics for injection +/- Azithromycin for Injection as initial treatment.
5. Signed informed consent form.

Exclusion Criteria:

Patients who meet any of the following criteria will not be included in the study:

1. Pneumonia is aquired more than 48h after admission or the patient was admitted to hospital within 30 days prior to admission.
2. Start antibiotic treatment before admission.
3. Gestational period or suckling period.
4. Admitted to ICU.
5. Immunocompromised patients.
6. Pneumonia is the terminal event of a serious disease.
7. Tuberculosis, lung cancer, non-infectious interstitial lung disease, pulmonary edema, atelectasis, pulmonary embolism, pulmanory eosinophilia, pulmonary vasculitis.
8. Allergic to the antibiotics of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients in the 17 centers of the study who meet the inclusion and exclusion criteria will be included.
Sampling Method: Probability Sample
Enrollment: 314 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-08-31 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
early deterioration or progression rate | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Xuezhong Yu, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Jun Xu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No